CLINICAL TRIAL: NCT01723878
Title: Observational, Post-authorization, Prospective Study for Evaluating Patterns of Disease Progression in Patients With Advanced Non-small-cell Lung Carcinoma (NSCLC) Harbouring EGFR Activating Mutations Treated With Erlotinib in First Line.
Brief Title: ASPET Study: An Observational Study of Tarceva (Erlotinib) in First Line in Patients With Advanced Non-Small Cell Lung Cancer Harbouring EGFR Activating Mutations
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28361
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the patterns of disease progression in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harbouring EGFR activating mutations receiving Tarceva (erlotinib) as first-line treatment. Patients will be followed for up to 12 months after progression of disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed locally advanced or metastatic (IIIB/IV) non-squamous non-small cell lung cancer (NSCLC) which is routinely evaluated in clinical practice according to RECIST criteria
* EGFR mutation-positive disease according to local laboratory testing
* Patients on treatment with Tarceva monotherapy as first-line treatment according to the physician's usual practice

Exclusion Criteria:

* Prior systemic therapy for advanced NSCLC. The administration of neoadjuvant or adjuvant chemotherapy is allowed as long as it was finalized >6 months prior to receiving Tarceva
* Participation in another clinical study
* Patients could have received radiotherapy as long as the irradiated lesion was not the only lesion for evaluating response and a long as the radiotherapy was completed before initiating Tarceva treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced non-small cell lung cancer (NSCLC) with EGFR activating mutations receiving first-line treatment with Tarceva
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2013-12-30 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (time from initiation of treatment to disease progression or death of any cause) in correlation with localization of progression and clinical tumor characteristics | 3 years

SECONDARY OUTCOMES:
Objective response rate, tumor assessments according to RECIST v1.1 criteria | 3 years
One-year overall survival (from initiation of treatment to 12 months after disease progression) | 3 years
Time to progression | 3 years
Exposure (dosage/duration) with first-line Tarceva in clinical practice | 3 years
Safety: Incidence of adverse events | 3 years
Velocity of progression (disease flares) after cessation of treatment with Tarceva following disease progression | 3 years
Treatments used after disease progression in clinical practice | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (43):
- Spain (43):
  - Hospital Virgen de los Lirios; Servicio de Oncologia, Alcoy, Alicante
  - Hospital Universitario Son Espases; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital General de Granollers; Servicio de Oncologia, Granollers, Barcelona
  - Hospital Mutua de Terrassa; Servicio de Oncologia, Terrassa, Barcelona
  - Hospital Universitario Puerta del Mar; Servicio de Oncologia, Cadiz, Cadiz
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Hospital de Donostia; Servicio de Oncologia Medica, Donostia / San Sebastian, Guipuzcoa
  - Hospital Infanta Sofia; Servico de Oncologia, San Sebastián de los Reyes, Guipuzcoa
  - Hospital General de Lanzarote, Lanzarote, Las Palmas
  - Hospital de Gran Canaria Dr. Negrin; Servicio de Oncologia, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Principe de Asturias; Servicio de Oncologia, Alcalá de Henares, Madrid
  - Fundacion Hospital de Alcorcon; Servicio de Oncologia, Alcorcón, Madrid
  - Hospital del Henares; Servicio de Oncologia, Coslada, Madrid
  - Complejo Hospitalario de Orense; Servicio de Oncologia, Ourense, Orense
  - Hospital Meixoeiro, Vigo, Pontevedra
  - Hospital Univ. Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias (HUC), La Laguna (Tenerife), Tenerife
  - Complejo Hospitalario Nuestra Señora de la Candelaria; Servicio de Oncologia, Santa Cruz de Tenerife, Tenerife
  - Hospital de Sagunto; Servicio de Oncologia, Sagunto, Valencia
  - Hospital Lluis Alcanys; Servicio de Oncologia, Xàtiva, Valencia
  - Hospital de Cruces; Servicio de Oncologia, Barakaldo, Vizcaya
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba
  - Hospital Universitario San Cecilio; Servicio de Oncologia, Granada
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Complejo Asistencial Universitario de Leon; Servicio de Oncologia, León
  - Complejo Hospitalario Xeral-Cies, Lugo
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Madrid
  - Hospital Universitario de Mostoles;Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Hematologia, Málaga
  - Hospital Universitario Virgen de Arrixaca; Servicio de Oncologia, Murcia
  - Hospital Clinico Universitario de Salamanca; Servicio de Oncologia, Salamanca
  - Hospital General de Segovia; Servicio de Oncologia, Segovia
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital General de Teruel Obispo Polanco; Servicio Oncologia, Teruel
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
  - Hospital Universitario Dr. Peset; Servicio de Oncologia, Valencia
  - Hospital Clinico Universitario de Valladolid; Servicio de Oncologia, Valladolid
  - Complejo Hospitalario Zamora- H. Virgen de la Concha; Servicio Oncologia, Zamora
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza